CLINICAL TRIAL: NCT06255314
Title: Evaluation of Minimally Invasive Ventral Hernioplasty With Extraperitoneal Mesh Placement
Brief Title: Minimally Invasive Techniques in Ventral Hernioplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Mohamed Badr, teaching assistant, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: laparoscopic ventral hernia
Record Dates: First submitted 2024-01-20; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- trans abdominal retromusclar laparoscopic ventral hernia repar (Experimental)
  Interventions: Procedure: ventral hernia repair
- enhanced view totally extraperitoneal laparoscopic ventral hernia repair (Experimental)
  Interventions: Procedure: ventral hernia repair
- open sublay ventral hernia repair (Experimental)
  Interventions: Procedure: ventral hernia repair

INTERVENTIONS:
Procedure: ventral hernia repair — Laparoscopic transabdominal retromuscular repair is a minimally invasive approach to the open Rives Stoppa retromuscular sublay repair for ventral hernia.
  In ventral hernia repair, it relies on initiation of dissection in one retrorectus space and then crossover to the contralateral retrorectus space The sublay mesh technique is an open surgical procedure for ventral and incisional hernias

SUMMARY:
1. Review the surgical outcome of different techniques using extraperitoneal ventral hernia repair regarding postoperative pain. wound infection ,hospital stay , recurrence ,mesh migration and mesh induced visceral complications.
2. Reviewing advantages and drawbacks of each surgical technique regarding feasibility ,cost effectiveness and technical difficulties

DETAILED DESCRIPTION:
The laparoscopic ventral hernia repair was first introduced by LeBlanc and Booth in the early 1990s . Since its introduction, it has continued to evolve and has become an important option in the hernia surgeon's armamentarium. However, only 27.4% of ventral hernia repairs are performed laparoscopically, likely because of the relatively advanced nature of this procedure and because all hernias may not be suitable for a laparoscopic approach. Using current techniques, numerous studies have documented the safety and efficacy of this approach. Some data suggest that the laparoscopic approach results in a shorter hospital stay and lower recurrence rates compared with open approaches. However, pain may still be significant after laparoscopic repairs and there are not significant advantages from this standpoint. Nonetheless, it is well accepted that the primary advantage of the laparoscopic approach is that wound infections are less frequent compared with open approaches .LeBlanc and Booth in 1993 first reported application of intra-peritoneal onlay mesh (IPOM) for ventral and incisional hernia, However the technique requires expensive fixation devices which may cause acute and chronic pain .The laparoscopic groin hernia repair using synthetic mesh in TEP or TAPP are acceptable surgical techniques today These techniques are rarely associated with mesh induced complications, the reason being extraperitoneal placement of synthetic mesh. It is apparent that despite great progress in mesh technology, nearly all types of meshes have been found to produce a varying level of adhesion or tissue reaction, regardless of the material and coating used. Preoperatively unpredictable, a mesh-induced visceral complication may occur in some patients to produce severe reaction or major mesh-related adverse events.The incitation to develop certain novel minimally invasive techniques that enables researchers to bring the mesh out of abdominal cavity has been an exciting trend in laparoscopic hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* • Able to give informed consent for inclusion in the study

  * Age of the patient : above 18 years
  * Any type of ventral hernia including umbilical,paraumbilical,epigastric,spigelian and incisional hernias

Exclusion Criteria:

* • Patients with inguinal hernia.

  * Strangulated or obstructed hernia.
  * Previous mesh hernia repair.
  * Loss of abdominal domain.
  * Infected or contaminated field.
  * Defect size more than 10cm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Operative time | from inflation of abdomen till deflation in laparoscopic repair and from skin incision up to skin closure in open repair.
Intra operative injuries including bowel or vascular injuries | intra operative

SECONDARY OUTCOMES:
• Surgical site infection | postoperative up to 1month
• Surgical site occurrence of hematoma ,seroma, necrosis | : 30 days
• Hernia recurrence | : 1year
Cost effectiveness | : 6months
  cost of polyprolene mesh compared to composite mesh by egyptian pound
•Rate of mesh related complication such as bowel erosion | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LeBlanc KA, Booth WV. Laparoscopic repair of incisional abdominal hernias using expanded polytetrafluoroethylene: preliminary findings. Surg Laparosc Endosc. 1993 Feb;3(1):39-41. PMID 8258069
- [Background] Colavita PD, Tsirline VB, Belyansky I, Walters AL, Lincourt AE, Sing RF, Heniford BT. Prospective, long-term comparison of quality of life in laparoscopic versus open ventral hernia repair. Ann Surg. 2012 Nov;256(5):714-22; discussion 722-3. doi: 10.1097/SLA.0b013e3182734130. PMID 23095614
- [Background] Jin J, Rosen MJ. Laparoscopic versus open ventral hernia repair. Surg Clin North Am. 2008 Oct;88(5):1083-100, viii. doi: 10.1016/j.suc.2008.05.015. PMID 18790156
- [Background] Golani S, Middleton P. Long-term follow-up of laparoscopic total extraperitoneal (TEP) repair in inguinal hernia without mesh fixation. Hernia. 2017 Feb;21(1):37-43. doi: 10.1007/s10029-016-1558-7. Epub 2016 Dec 26. PMID 28025740
- [Background] Muschalla F, Schwarz J, Bittner R. Effectivity of laparoscopic inguinal hernia repair (TAPP) in daily clinical practice: early and long-term result. Surg Endosc. 2016 Nov;30(11):4985-4994. doi: 10.1007/s00464-016-4843-8. Epub 2016 Mar 16. PMID 26983436
- [Background] Tung KLM, Cheung HYS, Tang CN. Non-healing enterocutaneous fistula caused by mesh migration. ANZ J Surg. 2018 Jan;88(1-2):E73-E74. doi: 10.1111/ans.13253. Epub 2015 Aug 5. No abstract available. PMID 26246228